CLINICAL TRIAL: NCT05936645
Title: The Efficacy of a Temporary Sub-Placental Uterine Tourniquet in Minimizing Intraoperative Blood Loss in Management of Placenta Accreta Spectrum Disorder by a Retrograde Cesarean Hysterectomy (Bladder Last): A Prospective Randomized Controlled Clinical Trial
Brief Title: The Efficacy of a Temporary Sub-Placental Uterine Tourniquet in Minimizing Intraoperative Blood Loss in Management of Placenta Accreta Spectrum Disorder by a Retrograde Cesarean Hysterectomy (Bladder Last)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Eltawil, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MD-429-2022
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Placenta Accreta
Keywords: Placenta Accreta Spectrum; Tourniquet; Cesarean Hysterectomy; Bladder Last; Blood loss
MeSH Terms: conditions — Placenta Accreta; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet Group (Experimental): A temporary sub-placental uterine tourniquet will be temporarily applied before fetal extraction.
  Interventions: Procedure: A temporary sub-placental Uterine Tourniquet in management of Placenta Accreta Spectrum disorder by a retrograde cesarean hysterectomy (Bladder Last)
- Non-Tourniquet Group (Experimental): No tourniquet will be used in this arm.
  Interventions: Procedure: Retrograde cesarean hysterectomy (Bladder Last) for management of Placenta Accreta Spectrum disorder

INTERVENTIONS:
Procedure: A temporary sub-placental Uterine Tourniquet in management of Placenta Accreta Spectrum disorder by a retrograde cesarean hysterectomy (Bladder Last) — Comparing the use of a temporary sub-placental uterine tourniquet versus no tourniquet in reducing blood loss in patients with Placenta Accreta Spectrum disorder undergoing cesarean hysterectomy.
  Arms: Tourniquet Group
Procedure: Retrograde cesarean hysterectomy (Bladder Last) for management of Placenta Accreta Spectrum disorder — Comparing the use of a temporary sub-placental uterine tourniquet versus no tourniquet in reducing blood loss in patients with Placenta Accreta Spectrum disorder undergoing cesarean hysterectomy.
  Arms: Non-Tourniquet Group

SUMMARY:
This trial will study the role of a temporary tourniquet around the uterus to reduce blood loss in management of patients with abnormally implanted placenta who will undergo removal of the uterus.

DETAILED DESCRIPTION:
Patients included in this study were subjected to:

* All the cases will be operated upon by the same surgical team including the same leads surgeon for all cases.
* Written consent: will be obtained from all participants who are included in the study.
* Full History Taking Including: Name, age , Obstetric code , Menstrual history and last menstrual period , Medical history , Surgical history
* Thorough Clinical Examination: including the vital signs (temperature, blood pressure, pulse, and respiratory rate) as well as the patient's height to weight ratio (body mass index).
* Laboratory tests: performed including complete blood count, prothrombin time, prothrombin concentration, liver and kidney function tests. Cross-matching of packed red blood cell units will be arranged beforehand.
* Ultrasound:

A detailed second-level trans-abdominal and trans-vaginal ultrasound will be scheduled and conducted before the date of delivery, by a single operator in the department's Ultrasound Unit using a GE Voluson F8 ultrasound system (GE Healthcare, Zipf, Austria).

Trans-abdominal ultrasound will be done in a supine position with both a full and an empty bladder to document fetal biometry, estimated fetal weight, amniotic fluid index and to screen signs of placental invasion. These signs include on grayscale ultrasound, loss of clear zone, myometrial thinning, presence of placental lacunae, bladder wall interruption, placental bulge and focal exophytic mass; and on color Doppler imaging (CDI), uterovesical hypervascularity; subplacental hypervascularity; bridging vessels and placental lacunae feeder vessels. The placenta was recorded as 'low lying' when its edge was 0.5-2 cm from the internal os of the uterine cervix on trans-vaginal ultrasound. When the placenta was < 0.5 cm from the internal os or completely covering it, it was defined as placenta previa (marginal or complete)

* At all-time the patient is closely monitored for hemodynamic instability or vaginal bleeding
* Patient positioning: the patient will be placed in the dorsal supine position
* A wide transverse incision will be performed.
* The rectus fascia and muscle are cut transversely and extended as far laterally as needed. The inferior epigastric vessels are identified and ligated bilaterally.
* The placental invasion will then be re-assessed.
* A partial bladder takedown will be performed to avoid inadvertent laceration of the placenta. This will be done by dissection and release of the adherent bladder from the anterior uterine wall as low as possible (utero-vesical peritoneal fold) together with the vascular disconnection of the newly formed vessels connecting the adherent invasive placenta to the urinary bladder.
* Tourniquet Group: A Foley catheter (20Fr) will be applied around the lower uterine segment at level lower than the placenta acting as a tourniquet
* The dissection of the utero-vesical fold will be extended laterally to both broad ligaments and bilateral opening in the anterior leaflet of the broad ligament will be made. Both ureters will be identified beforehand.
* A Foley catheter will be passed through the posterior leaflet of the left broad ligament in an avascular area , then passing the catheter back through the pouch of Douglas through the right broad ligament.
* The Foley catheter tourniquet will include both the lower uterine segment and part of the bladder dome.
* A Trans-vaginal ultrasound will be used intra-operatively to confirm the proper level of the tourniquet in all. Once the tourniquet is confirmed to be in a level below the placenta, the Foley catheter will be tightened and tied.
* A supra-placental hysterotomy incision is carried out immediately after tightening the tourniquet followed by fetal extraction with immediate cord clamping (< 30 seconds).
* The uterus is then exteriorized, kept under upward traction so that uterine vascular constriction can diminish blood loss and the hysterotomy incision bleeding is temporarily controlled by towel clips.
* We will wait for 10 minutes to assess placenta separation. We will proceed with the hysterectomy in a technique similar to the radical retrograde approach used for en-bloc resection of extensive pelvic disease.
* The round ligaments are divided and ligated, and the broad ligaments are incised laterally and parallel to the infundibulo-pelvic ligaments to expose the retroperitoneum. The loose areolar tissue encountered in this space is carefully dissected parallel to the ureters and the pelvic sidewall vessels.
* The utero-ovarian ligaments and tubes are divided and ligated bilaterally.
* The ureters are carefully identified, dissected and preserved through the anterior bladder pillar in order to keep them out of the field of dissection.
* The plane between the cervix and the bladder is identified below the tourniquet and careful dissection is performed
* The cervix is seized and pulled up behind the uterus. The retrograde approach is continued by retracting the uterus sharply upward, exposing the remaining cardinal ligament attachments (with uterine vessels) medial to the ureters, uterosacral ligaments and bladder pillars, which are sequentially divided by clamps and secured with suture ligatures.
* The uterine specimen removed is partially adherent to the bladder dome and is gently peeled off the bladder to avoid bladder injury with adequate control of the bridging vessels.
* The uterine stump is closed in 2 layers by continuous absorbable sutures.
* The temporary tourniquet is loosened to check for bleeding from the uterine stump and the back of the bladder. The tourniquet is then tightened again to temporarily control the bleeding.
* Individual bleeders from the back of the bladder are controlled by a right angle forceps and then suture ligated.
* Bleeding from the uterine stump is controlled by hemostatic sutures and electro-cautery.
* The tourniquet will be removed.
* Careful exploration is performed and adequate hemostasis is ensured
* Closure of the abdomen over 2 wide bore drains
* Non-Tourniquet group: (No tourniquet is applied around the lower uterine segment)
* Same technique without adding a temporary tourniquet around the uterine artery.
* Estimation of intraoperative blood loss will be obtained through measuring the volume of blood in the suction machine reservoir and weighing the swabs (surgical towels) as soon as possible. The weights of dry swabs will be subtracted from the weights of swabs used during the operation. The weight of swabs found in grams will be translated to ml by using blood density (1.050 g/ml)
* Postoperative blood loss in the first 24 hours and after will be measured by subtracting intraoperative blood loss from the total blood loss
* For patients who didn't receive intra-operative or post-operative blood transfusion, total blood loss will be measured through pre and post operative hematocrit values through the following equations:

The estimated total blood loss will be derived by multiplying the calculated pregnancy blood volume by percentage of blood volume lost.

Pregnancy blood volume = (0.75 × {[maternal height (inches) × 50] + [maternal weight in pounds × 25]}) Percent of blood volume lost = ({predelivery Hematocrit - postdelivery hematocrit}/pre-delivery hematocrit)

Total blood loss = pregnancy blood volume × percent of blood volume lost - The need for blood transfusion and its amount intra or post-operative will be recorded

- For patients who had intra or postoperative blood transfusion, the actual blood loss was calculated through Lopez-Picado's formula: Estimated blood loss (m) = [Estimated blood volume x (pre-operative hematocrit-post-operative hematocrit) + vol. of transfused packed red blood cells]/average hematocrit Where Average hematocrit is the sum of preoperative & postoperative hematocrit levels, divided by 2.

According to the International Council for Standardization in Hematology (ICSH):

For women: Estimated blood volume (EBV) (ml) = Plasma vol. (ml) + Red cell vol. (ml) = [weight (kg) ^0.425 × height (cm) ^0.725 x 0.007184 x2.217] + [age(years) x1.061]

* Pre and 24-h post-operative hemoglobin (g/dl).
* Operative time and post-operative hospital stay will be recorded.
* Close post-operative monitoring of the patients' vital signs, drain output and urine output
* Presence or absence of intraoperative complications; bladder, ureteric, bowel or vascular injuries will be recorded.
* Monitoring for post-operative morbidities as postpartum hemorrhage, DVT, claudications, or the need for ICU admission, all will be recorded.
* Randomization: The 30 included participants will be subjected to block randomization into 5 blocks containing 6 participants each by a single member of the research team.

  * The participants will be assigned into the blocks by chronological order on the day prior to the operation.
  * The outcome of the randomization process will be concealed from the patients.
  * The surgical team will be informed about the outcome of the randomization process for each patient on the day of the operation.
  * T stands for the tourniquet group while N stands for the non-tourniquet group

Block 1 TNNTTN Block 2 TTNNNT Block 3 NTNNTT Block 4 NNTNTT Block 5 TNTNTN

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: pregnancy completing 35 weeks or more.
* Previous one or more cesarean delivery.
* Current pregnancy complicated by Placenta Accreta Spectrum Disorder candidate for cesarean hysterectomy either total or partial Placenta Accreta. (i.e. Total: Most of the placenta is adherent to the myometrium with no plane of cleavage. Partial: 2-3 cotyledons are only adherent to the myometrium with no plane of cleavage at these cotyledons)
* Elective termination of pregnancy.
* Preoperative Hemoglobin ≥ 10 g/dl

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Women with history of a concomitant chronic or a pregnancy associated medical disorder eg. Gestational diabetes, hypertension, cardiac or renal disease.
* Presence of a concomitant uterine pathology (eg. Uterine fibroid)
* Premature rupture of membranes.
* Cases misdiagnosed as placenta accreta by ultrasound preoperatively, and spontaneous full placental separation occurred intraoperative or as total/partial accreta and found to be focal accreta intraoperative.
* Cases requiring preoperative blood transfusion.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
The estimated total blood loss. | 24 hours
  ml

SECONDARY OUTCOMES:
Operative time | From the start of the procedure till the end.
  minutes
Need for blood transfusion | before, during and immediately after the procedure
  Number of units of packed blood transfused
Internal organ injury (Bladder, intestine, ureter) | during the operative procedure
  Injury to bladder, intestine or ureter
Inadvertent injury to the pelvic vessels (eg. Injury to the ovarian vessels while inserting the tourniquet) | during the operative procedure
  Injury to major pelvic vessel
ICU admission | immediately after the procedure
  post operative ICU admission
Neonatal APGAR score | at 1 and 5 minutes after birth
  APGAR (Appearance, Pulse, Grimace, Activity and Respiration) score of the newborn. The score is scaled from 0 to 10, where a higher score indicates a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Moutaz M Elsherbini, MD, Study Director — Department of Obstetrics and Gynecology, Faculty of Medicine, Cairo University, Cairo, Egypt
Locations (1):
- Research Ethics Committee, Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data related to the published results after deidentification (texts, tables, figures and appendices)
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication and no end date
Access Criteria: anyone who wishes to access the data

REFERENCES:
- [Background] Alves ALL, Silva LBD, Costa FDS, Rezende GC. Management of placenta accreta spectrum. Rev Bras Ginecol Obstet. 2021 Sep;43(9):713-723. doi: 10.1055/s-0041-1736371. Epub 2021 Oct 20. No abstract available. PMID 34670307
- [Background] Altal OF, Qudsieh S, Ben-Sadon A, Hatamleh A, Bataineh A, Halalsheh O, Amarin Z. Cervical tourniquet during cesarean section to reduce bleeding in morbidly adherent placenta: a pilot study. Future Sci OA. 2022 Mar 8;8(4):FSO789. doi: 10.2144/fsoa-2021-0087. eCollection 2022 Apr. PMID 35369280
- [Background] Bartels HC, Postle JD, Downey P, Brennan DJ. Placenta Accreta Spectrum: A Review of Pathology, Molecular Biology, and Biomarkers. Dis Markers. 2018 Jul 3;2018:1507674. doi: 10.1155/2018/1507674. eCollection 2018. PMID 30057649
- [Background] Donovan BM, Shainker SA. Placenta Accreta Spectrum. Neoreviews. 2021 Nov;22(11):e722-e733. doi: 10.1542/neo.22-11-e722. PMID 34725137
- [Background] Huang J, Zhang X, Liu L, Duan S, Pei C, Zhao Y, Liu R, Wang W, Jian Y, Liu Y, Liu H, Wu X, Zhang W. Placenta Accreta Spectrum Outcomes Using Tourniquet and Forceps for Vascular Control. Front Med (Lausanne). 2021 Oct 18;8:557678. doi: 10.3389/fmed.2021.557678. eCollection 2021. PMID 34733857
- [Background] Hussein AM, Elbarmelgy RA, Elbarmelgy RM, Thabet MM, Jauniaux E. Prospective evaluation of impact of post-Cesarean section uterine scarring in perinatal diagnosis of placenta accreta spectrum disorder. Ultrasound Obstet Gynecol. 2022 Apr;59(4):474-482. doi: 10.1002/uog.23732. Epub 2022 Mar 8. PMID 34225385
- [Background] Jauniaux E, Hussein AM, Elbarmelgy RM, Elbarmelgy RA, Burton GJ. Failure of placental detachment in accreta placentation is associated with excessive fibrinoid deposition at the utero-placental interface. Am J Obstet Gynecol. 2022 Feb;226(2):243.e1-243.e10. doi: 10.1016/j.ajog.2021.08.026. Epub 2021 Aug 28. PMID 34461077
- [Background] Morlando M, Collins S. Placenta Accreta Spectrum Disorders: Challenges, Risks, and Management Strategies. Int J Womens Health. 2020 Nov 10;12:1033-1045. doi: 10.2147/IJWH.S224191. eCollection 2020. PMID 33204176
- [Background] Stafford I, Dildy GA, Clark SL, Belfort MA. Visually estimated and calculated blood loss in vaginal and cesarean delivery. Am J Obstet Gynecol. 2008 Nov;199(5):519.e1-7. doi: 10.1016/j.ajog.2008.04.049. Epub 2008 Jul 17. PMID 18639209